CLINICAL TRIAL: NCT05528224
Title: Effect of Stepped Care in Internet-Based Cognitive Behavioral Therapy for Adults With Obsessive-Compulsive Disorder：A Three-Arm Randomized Controlled Trial
Brief Title: Effect of SC-ICBT for Adults With OCD：A Three-Arm Randomized Controlled Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Main trial terminated after pilot trial: full randomization proved infeasible for nonlocal participants; baseline symptom-based allocation added confounding variable; comparison with CBGT alone was deemed sufficient to assess SC-ICBT effectiveness
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OCDICBT2022-36
Record Dates: First submitted 2022-08-11; First posted 2022-09-06 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Obsessive-Compulsive Disorder; Stepped-care Internet-based Cognitive Behavioral Therapy; Cost-effectiveness; Randomized Controlled Trial
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- stepped-care Internet-based cognitive behavioral therapy(SC-ICBT) combined with medication (Experimental): In the main study, after individualized assessment（0 week and 3 week separately）, OCD patients will be provided with self-guided ICBT or therapist-guided ICBT through the severity of their symptoms flexibly while they will continue with the medications they already have.
  In the pilot study, 23 OCD patients will be assigned to SC-ICBT group based on their autonomous will. They will begin with self-guided ICBT, followed by an assessment of their treatment outcomes at week 3, with non-responders being escalated to a higher intensity of treatment, and additional therapist-guided ICBT in the following three weeks. During the 6-week treatment they will continue with the medications they already have.
  Interventions: Other: stepped-care Internet-based cognitive behavioral therapy(SC-ICBT); Drug: conventional medical treatment (TAU)
- Cognitive Behavioral Group Therapy (CBGT) combined with medication (Active Comparator): In the main study, OCD patients will be provided with therapist-guided offline Cognitive Behavioral Group Therapy while they will continue with the medications they already have.
  In the pilot study, 23 OCD patients will be assigned to CBGT group based on their autonomous will. They will receive the same CBGT intervention as in the main study while they will continue with the medications they already have.
  Interventions: Other: Cognitive Behavioral Group Therapy (CBGT); Drug: conventional medical treatment (TAU)
- conventional medical treatment (TAU) (Active Comparator): In the main study, OCD patients will be treated as usual. Namely, they will continue with the medications they already have.
  This group is not present in the pilot study, as both SC-ICBT group and CBGT group combines medications. We suppose that the mere use of SC-ICBT group compared to CBGT group (a commonly used psychotherapy in Chinese clinical practice) is sufficient to draw conclusions about the feasibility of SC-ICBT in in adults with OCD in China.
  However, in order to further validate the economic benefits of SC-ICBT, we chose to set TAU group in the main study.
  Interventions: Drug: conventional medical treatment (TAU)

INTERVENTIONS:
Other: stepped-care Internet-based cognitive behavioral therapy(SC-ICBT) — OCD patients will take part in four structured online lessons for 6 weeks. Lesson one: Psychological Health Education, including the knowledge about OCD, SUDs and other related information.
  Lesson two: Exposure and Response Prevention (ERP), including the knowledge about ERP, exposure item list and other related information.
  Lesson three: Practice of Exposure and Response Prevention. Patients are asked to perform ERP practice based on what they have learned previously: practice at least once a day, a day about one hour all together. On this basis, in the main study, patients with severe obsessive and compulsive symptoms(Y-BOCS≥24) will be provided with extra therapist-guided ICBT: twice a week, about an hour one time. While in the pilot study, non-responders at week 3(YBOCS score reduction rate<25%) will be provided with extra therapist-guided ICBT.
  Lesson four: Practice retrospection and relapse prevention.
  Arms: stepped-care Internet-based cognitive behavioral therapy(SC-ICBT) combined with medication
Other: Cognitive Behavioral Group Therapy (CBGT) — OCD patients will be asked to come to Shanghai Mental Health Center to take part in the offline CBT group. Each group will be treated for 6 weeks, twice a week for 2 hours each time. The treatment was supervised by an experienced CBGT therapist. The structure of the course basically corresponds with the SC-ICBT group.
  Arms: Cognitive Behavioral Group Therapy (CBGT) combined with medication
Drug: conventional medical treatment (TAU) — In this study, the investigators use selective serotonin reuptake inhibitors (SSRIs) approved by the State Food and Drug Administration (CFDA) for the treatment of OCD (i.e., fluoxetine, paroxetine, sertraline and fluvoxamine) as well as citalopram and escitalopram. The second-generation atypical antipsychotics may also be combined as a potentiator if the patient requires.
  The maximum dosage shall not exceed the maximum dosage prescribed in the instruction manual.

SUMMARY:
The goal of this clinical trial is to learn about the efficacy and cost-effectiveness of stepped-care Internet-based cognitive behavioral therapy (SC-ICBT) compared with Cognitive Behavioral Group Therapy (CBGT) and conventional medical treatment (treatment as usual, TAU) in adults with obsessive-compulsive disorder (OCD) in China.

The main questions it aims to answer are:

question 1: Whether the efficacy of SC-ICBT is noninferior to CBGT and TAU for OCD?

question 2: Whether SC-ICBT is more cost-effective than CBGT and TAU for OCD?

Participants will receive treatment (SC-ICBT or CBGT or TAU) for 6 weeks.

Prior to the main study, we conduct a non-randomized pilot study to explore the efficacy and cost-effectiveness of SC-ICBT related to CBGT for adults with OCD in China.

DETAILED DESCRIPTION:
Internet-based cognitive behavioral therapy (ICBT) integrates the Internet and cognitive behavioral therapy, which enables patients to participate in different treatment modules online. ICBT has been proved to be an effective way to improve the symptoms of OCD patients with lower cost. Stepped care model (SCM) allows to better balance the efficacy of treatment and the cost of treatment.

In the main study, the investigators plan to develop an intervention pattern of stepped-care Internet-Based cognitive behavioral therapy (SC-ICBT): After individualized assessment（0 week and 3 week separately）, OCD patients will be provided with self-guided ICBT or therapist-guided ICBT through the severity of their symptoms flexibly. This study will be a randomized, controlled, assessor-blinded trial of three groups in OCD: Stepped-care Internet-based Cognitive Behavioral Therapy (SC-ICBT) combined with medication, Cognitive Behavioral Group Therapy (CBGT) combined with medication, and conventional medical treatment (TAU). The study aims to investigate the efficacy and cost-effectiveness of SC-ICBT related to CBGT and TAU for adults with OCD in China.

To initially validate the feasibility of SC-ICBT in Chinese patients with OCD, the investigators plan to firstly conduct a small, non-randomized pilot study prior to the main study. In the pilot study, patients assigned to SC-ICBT group will begin with self-guided ICBT, followed by an assessment of their treatment outcomes at week 3, with non-responders being escalated to a higher intensity of treatment, and additional therapist-guided ICBT in the following three weeks.

In the main study, the investigators plan to recruit 114 OCD patients and randomly assigns them to the SC-ICBT group, CBGT group, and TAU group for treatment of 6 weeks and follow-up of 3 months.

While in the pilot study, 46 OCD patients will be recruited and assigned to the SC-ICBT group or CBGT group based on their autonomous will.

Questionnaires, scales, behavior experiments and other experimental materials will be used to evaluate the intervention effect of 6-week SC-ICBT on obsessive and compulsive symptoms, cognitive function and quality of life of OCD patients as well as patients' and therapists' cost.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 50 years
2. Satisfied with the diagnostic criteria for OCD in DSM-5.
3. 16≤YBOCS score ≤31
4. Taking medication stably for 8 weeks
5. Education level ⩾6 years
6. Has sufficient audiovisual skills to complete the necessary examinations for the study.
7. Right-handed (this criterion is for fMRI subjects only)
8. Subjects and their guardians understood the study and signed informed consent.

Exclusion Criteria:

1. Satisfied with the diagnostic criteria for a mental disorder in DSM-V other than OCD.
2. Obsessive-compulsive symptoms were too severe to participate in the experiment.
3. High risk of suicide.
4. Severe central system or physical disease
5. Pregnant women or women that getting ready for being pregnant and lactating.
6. Other treatments being performed.
7. Uncooperative or unable to complete treatment
8. With metal implants in the body, such as pacemakers, intracranial silver clips, metal dentures, arterial stents, arterial clips, joint metal fixation, or other metal implants, etc. (this criterion is for fMRI subjects only)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Change of Yale-Brown Obsessive-Compulsive Scale (YBOCS) | Change from Baseline at 6weeks
  YBOCS is compiled by Goodman in the United States and contains 10 items to assess the severity of obsessive thoughts and compulsive behavior. The scoring method adopts a five-point scale of 0-4 points, and the total score range is 0-40 points, which has good reliability and validity.

SECONDARY OUTCOMES:
Change of Florida Obsessive-Compulsive Inventory (FOCI) | Change from Baseline at 6weeks
  FOCI, a self-rating scale, is used to assess the severity of obsessive-compulsive symptoms within one month, which contains 20 items. The first 15 items are evaluated the symptoms by yes and no, and the last 5 items are evaluated the severity of symptoms on 0-4 five-point scale.
Change of Self-rating Depression Scale (SDS) | Change from Baseline at 6weeks
  Self-rating Depression Scale (SDS) was developed by William W. K. Zung of Duke University Medical School in 1965. It is one of the most widely used self-rating depression scales. It is used to measure the severity of depression and its change in treatment.
Change of Self-rating Anxiety Scale (SAS) | Change from Baseline at 6weeks
  The Self-rating Anxiety Scale (SAS) is very similar to the Self-rating Depression Scale (SDS) from the scale construction to the evaluation method. It is a very simple clinical tool to analyze the subjective anxiety symptoms of patients. It is suitable for adults with anxiety symptoms and has a wide range of application.

OTHER OUTCOMES:
Change of 36-item Short Form Health Survey（SF-36） | Change from Baseline at 6weeks
  36-item Short Form Health Survey（SF-36）will be used to assess the health-related quality of life of patients. SF-36 is one of the most commonly used standardized measurement tools for quality of life in the world, including eight subscales, a total of 36 items, involving physical and mental health.
Cost-effectiveness analysis | the cost from Baseline to Week 6
  The study designs a self-rated questionnaire about cost-effectiveness analyses, including both direct and indirect costs, and the patients themselves fill out the questionnaire based on the bill.
  The cost-effectiveness analysis method (CEA) is used to measure the spending of three groups. The results of the total cost divided by YBOCS total reduction scores can reflect the cost required to obtain each unit of curative effect.
Cost-utility analysis | the cost from Baseline to Week 6
  The cost-utility analysis method is used to measure the spending of improving patients' quality of life. The results of the total cost divided by SF-36 total improvement scores can reflect the cost required to obtain each unit of utility.
Dropout rate | From Baseline to Week 6
  Dropout rate is recorded to evaluate treatment acceptability.
Frequency of occurrence | From Baseline to Week 6
  Frequency of occurrence is recorded to evaluate treatment acceptability. The investigators use sign-in sheets to measure patients' attendance during the treatment.
Homework completion | From Baseline to Week 6
  Homework completion is recorded to evaluate treatment acceptability. The investigators use sign-in sheets to keep track of patients' homework completion.
Subjective satisfaction with treatment | From Baseline to Week 6
  Subjective satisfaction with treatment is recorded to evaluate treatment acceptability. The investigators use a self-rated question（"Overall, how satisfied are you with your current treatment?") to measure patients' subjective satisfaction. The rating was done on a 7-item scale ranging from "Extremely dissatisfied" to "Extremely satisfied".
Treatment safety | From Baseline to Week 6
  Adverse events (AEs) are the treatment safety indicators
Change of randomized dot motion(RDM) perceptual decision-making task | Change from Baseline at 6weeks
  RDM is a classical perceptual decision paradigm, in which subjects need to report the overall movement direction of 300 randomly moving white dots, and the total duration of the task is about 25 minutes. RDM is often used together with drift diffusion models to study human decision-making processes and has been supported by many research evidences. After the RDM decision, a confidence assessment stage is added to measure the decision confidence of the subjects through their subjective reports.
Change of the antisaccade task | Change from Baseline at 6weeks
  The antisaccade task is a classical experimental paradigm to measure the response inhibition ability of subjects in the field of cognitive function.
Change of the task-state functional magnetic resonance imaging(fMRI) of the whole brain | Change from Baseline at 6weeks
  The investigators use the randomized dot motion perceptual decision-making task as Neuroimaging Paradigm to observe the neurophysiological changes cauesd by step-ICBT in patients with OCD.

CONTACTS AND LOCATIONS:
Overall Officials: Qing Fan, Doctor, Study Chair — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China